CLINICAL TRIAL: NCT00424801
Title: Intensive Non-Sympathetic Activating Vasodilatory Treatment in Hypertensive Patients With Microvascular Angina Pectoris
Brief Title: Effects of Intensive Long-Term Vasodilation in Hypertensive Patients With Microvascular Angina Pectoris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to recent findings relating MRI contrast to nephrogenic systemic fibrosis
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cardiovascular Research Academy (Unknown); Danish Heart Foundation (Other); Novartis (Industry)
Responsible Party: Kent Lodberg Christensen, DMSc, Aarhus Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vasointense
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Microvascular Angina; Hypertension
MeSH Terms: conditions — Microvascular Angina; Hypertension | interventions — lercanidipine; Valsartan; Nicorandil; Doxazosin; moxonidine; Pindolol; amiloride, hydrochlorothiazide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vasodilatory (Experimental): Patients in this arm will receive intensive vasodilatory treatment to lower blood pressure
  Interventions: Drug: Lercanidipine; Drug: Valsartan; Drug: Nicorandil; Drug: Doxazosin; Drug: Moxonidin; Drug: Pindolol; Drug: Amiloride, hydrochlorothiazide

INTERVENTIONS:
Drug: Lercanidipine — Individual titration, max. dose 20 mg OD for 8 months
  Other Names: Zanidip
Drug: Valsartan — Individual titration, max. dose 160 mg OD for 8 months
  Other Names: Diovan
Drug: Nicorandil — Individual titration, max. dose 20 mg BD for 8 months
  Other Names: Angicor
Drug: Doxazosin — Individual titration, max. dose 4 mg OD for 8 months
  Other Names: Doxazosin "Stada"
Drug: Moxonidin — Possible add-on therapy in case target blood pressure can not be reached with a combination of the other drugs in the Vasodilatory arm. Individual titration, max. dose 0,2 mg OD for 8 months
  Other Names: Moxonidin "Alpharma"
Drug: Pindolol — Possible add-on therapy in case target blood pressure can not be reached with a combination of the other drugs in the Vasodilatory arm. Individual titration, max. dose 10 mg OD for 8 months
  Other Names: Visken
Drug: Amiloride, hydrochlorothiazide — Possible add-on therapy in case target blood pressure can not be reached with a combination of the other drugs in the Vasodilatory arm. Individual titration, max. dose 1 tbl. OD for 8 months
  Other Names: Sparkal

SUMMARY:
The purpose of this study is to determine if long-term vasodilatory treatment is more effective than the standard treatment in hypertensive patients with microvascular angina pectoris

DETAILED DESCRIPTION:
Patients with hypertension frequently develop angina pectoris. This can be caused by either epicardial stenotic disease or, equally frequent, by increased resistance in small resistance vessels - microvascular dysfunction. This increased resistance is caused by a process called remodelling, where the existing material in the vessel wall is rearranged around a smaller lumen, whereas the sensitivity of the smooth muscle cells to agonist stimuli is unchanged. Under resting conditions the resistance is determined by both the tone in the smooth muscle cells in the vessel walls and the structure of the vessels themselves (RREST). Under hyperemic conditions the muscles relax and the resistance is determined only by vessel structure (RMIN).

A literature survey of the various studies on this subject has shown that structural changes relates to tone rather than blood pressure. This suggests that resistance vessel structure will be normalized only by an antihypertensive treatment which normalizes RREST i.e. rely on vasodilatation as a cause of the antihypertensive effect more than reduction of cardiac output.

The main hypothesis is, that it is possible to reverse the structural changes in the resistance vessels by vasodilatory treatment for eight months, thereby achieving lower coronary and peripheral minimal resistance (as determined by MRI and plethysmography, respectively), higher work capacity on exercise-ECG and less tendency to angina in these patients.

We will include 80 patients with essential hypertension, angina pectoris CCS class II-III and signs of ischemia on exercise-ECG or myocardial SPECT, but without significant stenosis in angiography. The patients are randomised, in a parallel, open-label design, to either vasodilatory (lercanidipine, valsartan, doxazosin and nicorandil) or standard treatment (metoprolol, diltiazem and isosorbide mononitrate). The aim of treatment in both arms is BP below 120/80 and the protocol allows further add-on therapy to reach this goal. The patients will be followed for eight months with a titration period of two months. MRI, plethysmography, exercise-ECG and echocardiography will be performed before and after the study period. The primary endpoint is minimal coronary resistance as determined by MRI; secondary endpoints are peripheral vascular resistance as determined by plethysmography, work capacity and ischemia threshold on exercise-ECG or myocardial SPECT.

ELIGIBILITY:
Inclusion Criteria:

* hypertension
* angina pectoris CCS class II-IV
* objective signs of ischemia on exercise-ECG or myocardial SPECT
* no significant stenosis on angiography (minimal lumen diameter >50% of relevant reference segment)

Exclusion Criteria:

* known allergy to any study medication
* abnormal lab tests of clinical significance
* valvular disease of haemodynamic significance
* known secondary hypertension
* atrial fibrillation or other significant arrythmias
* myocardial infarction < 30 days before inclusion
* resting angina < one week before inclusion
* known endocrine disease, nephropathy or hepatic disease
* present malignant disease
* pregnancy
* fertile women not using safe contraceptives > 6 months before inclusion. Use of contraceptives must continue 1 month after completion or retraction from the study
* body mass index > 30
* significant chronic obstructive lung disease (FEV1 < 1.5 l)
* participant in another study including test medicine
* present treatment with dipyridamole
* present treatment with phosphodiesterase-5-inhibitors that the patient does not want to discontinue during the study period
* heart transplanted patients
* patients with magnetizable metallic implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Minimal coronary resistance | 8 months

SECONDARY OUTCOMES:
Peripheral vascular resistance | 8 months
Work capacity | 8 months
Ischemia threshold | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Præstholm, MD, Principal Investigator — University of Aarhus; Kent L Christensen, MD, DrMSc, Study Director — Aarhus Hospital, medical-cardiologic dept. A; Won Yong Kim, MD, DrMSc, Study Director — Skejby Hospital, cardiologic dept. B; Hans Erik Bøtker, MD, DrMSc, Study Director — Skejby Hospital, cardiologic dept. B
Locations (1):
- Aarhus Hospital, Aarhus, Denmark